CLINICAL TRIAL: NCT02246777
Title: Assessment of Efficacy and Safety of the EX-PRESS® Glaucoma Filtration Device in Patients With Normal Tension Glaucoma
Brief Title: Alcon® Ex-PRESS® Glaucoma Filtration Device in Japanese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALJ-P2013-1; UMIN000013243 (Registry Identifier: UMIN)
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ex-PRESS (Experimental): Ex-PRESS® Glaucoma Filtration Device, Model P50PL, implanted in the anterior chamber of the study eye during glaucoma surgery intended for the lifetime of the patient
  Interventions: Device: Ex-PRESS® Glaucoma Filtration Device, Model P50PL

INTERVENTIONS:
Device: Ex-PRESS® Glaucoma Filtration Device, Model P50PL

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the Alcon Ex-PRESS® Glaucoma Filtration Device (Ex-PRESS) in Japanese subjects with normal tension glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of normal tension glaucoma.
* Indicated for filtration surgery using Ex-PRESS®.
* Understand and provide Informed Consent.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women who are pregnant, lactating, or planning to be pregnant during the study period.
* Diagnosis of angle closure glaucoma or secondary glaucoma.
* History of glaucoma surgery.
* Ophthalmologic surgery within the past 6 months.
* Difficulty with applanation tonometry measurement.
* Corneal dystrophy.
* Infectious/non-infectious conjunctivitis, keratitis, or uveitis in either eye.
* Severe blepharitis or dry eye.
* History of metal allergy.
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon Japan, Ltd.
Locations (1):
- Contact Alcon Japan, Ltd for Trial Locations, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 study centers located in Japan.
Period: Overall Study
Arm/Group | Ex-PRESS
Started | 32
Completed | 29
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Change of residence | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects after use of the investigational device (Safety Analysis Set).
Arm/Group | Ex-PRESS
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmHG] — IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Population: This analysis population includes all subjects treated with the investigational device, whose test/assessment data after the use of the device were available, having no inclusion/exclusion criteria violation substantially affecting the efficacy evaluation (Intent-to-Treat Analysis Set).
  mmHG
    number analyzed (Participants) | 29
    (all) | 14.8 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP)
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Only one eye contributed to the analysis.
Time Frame: Month 3, Month 6, Month 12 Post-Operative
Population: Intent-to-Treat, with non-missing data
Measure: Mean (Standard Deviation); unit: mmHG
Units Other Than Participants: Eyes
Arm/Group | Ex-PRESS
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 29
mmHG
  Month 3 | 9.4 (4.3)
  Month 6: number analyzed (Participants) | 28
  Month 6: number analyzed (Eyes) | 28
  Month 6 | 9.5 (3.8)
  Month 12: number analyzed (Participants) | 26
  Month 12: number analyzed (Eyes) | 26
  Month 12 | 10.0 (3.1)

2. Primary Outcome: Change From Baseline in IOP
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye contributed to the analysis.
Time Frame: Baseline (Pre-Operative), Month 3, Month 6, Month 12 Post-Operative
Population: Intent-to-Treat, with non-missing data
Measure: Mean (Standard Deviation); unit: mmHG
Units Other Than Participants: Eyes
Arm/Group | Ex-PRESS
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 29
mmHG
  Month 3 | -5.4 (4.6)
  Month 6: number analyzed (Participants) | 28
  Month 6: number analyzed (Eyes) | 28
  Month 6 | -5.4 (4.8)
  Month 12: number analyzed (Participants) | 26
  Month 12: number analyzed (Eyes) | 26
  Month 12 | -4.9 (4.2)

3. Primary Outcome: Percent Change From Baseline in IOP
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative percent change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye contributed to the analysis.
Time Frame: Baseline (Pre-Operative), Month 3, Month 6, Month 12 Post-Operative
Population: Intent-to-Treat, with non-missing data
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: Eyes
Arm/Group | Ex-PRESS
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 29
percent change
  Month 3 | -35.4 (30.1)
  Month 6: number analyzed (Participants) | 28
  Month 6: number analyzed (Eyes) | 28
  Month 6 | -33.7 (33.5)
  Month 12: number analyzed (Participants) | 26
  Month 12: number analyzed (Eyes) | 26
  Month 12 | -31.1 (23.6)

4. Primary Outcome: Percentage of Eyes With IOP Lowering Rate of 20% or More From Baseline up to Month 12
Description: as for outcome 1
Time Frame: Baseline (Pre-Operative), Month 3, Month 6, Month 12 Post-Operative
Population: Intent-to-Treat, with non-missing data
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Ex-PRESS
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 29
percentage of eyes
  Month 3 | 72.4
  Month 6: number analyzed (Participants) | 28
  Month 6: number analyzed (Eyes) | 28
  Month 6 | 82.1
  Month 12: number analyzed (Participants) | 26
  Month 12: number analyzed (Eyes) | 26
  Month 12 | 61.5

5. Primary Outcome: Percentage of Eyes Receiving Drug Therapy for Glaucoma Necessary to Maintain the IOP
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). For some subjects, both left and right eyes were targeted for the study, and data from both eyes were analyzed for this safety endpoint, as specified in the protocol.
Time Frame: Month 3, Month 6, Month 12 Post-Operative
Population: Intent-to-Treat Analysis Set with non-missing data
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Ex-PRESS
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 34
percentage of eyes
  Month 3 | 0.0
  Month 6: number analyzed (Participants) | 28
  Month 6: number analyzed (Eyes) | 33
  Month 6 | 0.0
  Month 12: number analyzed (Participants) | 26
  Month 12: number analyzed (Eyes) | 31
  Month 12 | 3.2

6. Primary Outcome: Percentage of Eyes Receiving Secondary Surgical Treatment (Including Laser Therapy) Necessary to Maintain the IOP
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Secondary surgical treatment included needling, laser suture lysis, and conjunctival and scleral flap sutures. For some subjects, both left and right eyes were targeted for the study, and data from both eyes were analyzed for this safety endpoint, as specified in the protocol. An eye may have received more than one procedure.
Time Frame: Month 3, Month 6, Month 12 Post-Operative
Population: Intent-to-Treat, with non-missing data
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Ex-PRESS None: No secondary surgical intervention
- Ex-PRESS + Needling: Ex-PRESS® Glaucoma Filtration Device with needling as a secondary surgical treatment
- Ex-PRESS + Laser Suture Lysis: Ex-PRESS® Glaucoma Filtration Device with laser suture lysis as a secondary surgical treatment
- Ex-PRESS + Conjunctival Suture: Ex-PRESS® Glaucoma Filtration Device with conjunctival suture as a secondary surgical treatment
- Ex-PRESS + Scleral Flap Suture: Ex-PRESS® Glaucoma Filtration Device with scleral flap suture as a secondary surgical treatment
Arm/Group | Ex-PRESS None | Ex-PRESS + Needling | Ex-PRESS + Laser Suture Lysis | Ex-PRESS + Conjunctival Suture | Ex-PRESS + Scleral Flap Suture
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
Number analyzed (Eyes) | 34 | 34 | 34 | 34 | 34
percentage of eyes
  Month 3 | 88 | 12 | 0 | 0 | 0
  Month 6: number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
  Month 6: number analyzed (Eyes) | 33 | 33 | 33 | 33 | 33
  Month 6 | 94 | 3 | 0 | 3 | 3
  Month 12: number analyzed (Participants) | 26 | 26 | 26 | 26 | 26
  Month 12: number analyzed (Eyes) | 31 | 31 | 31 | 31 | 31
  Month 12 | 100 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 15 months). This analysis population includes all subjects/eyes treated with the investigational device (32 subjects/37 eyes). Number at risk is reported in unit "eyes."
Description: An AE was defined as all undesirable or unintended signs, symptoms or diseases that occur from the start of the filtration surgery using Ex-PRESS®, regardless of the causal relationship with the filtration surgery using Ex-PRESS®. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Arm/Group | Ex-PRESS
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 13/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ex-PRESS (N=37)
Choroidal detachment (Eye disorders) | 5
Hyphaema (Eye disorders) | 4
Corneal epithelium defect (Eye disorders) | 2
Macular fibrosis (Eye disorders) | 1
Macular oedema (Eye disorders) | 1
Blebitis (Eye disorders) | 1
Optic disc haemorrhage (Eye disorders) | 1
Maculopathy (Eye disorders) | 1

LIMITATIONS AND CAVEATS:
This study was a single-arm study with filtration surgery using EX-PRESS®. Although target sample size was 45 patients, only 32 patients (37 eyes) were enrolled due to a small number of patients meeting eligibility criteria of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.